CLINICAL TRIAL: NCT05007275
Title: A Phase I Study to Determine Safety and Immunogenicity of the Candidate COVID-19 Vaccine AZD1222 Delivered by Aerosol in Healthy Adult Volunteers
Brief Title: A Study to Determine Safety and Immunogenicity of the Candidate COVID-19 Vaccine AZD1222 Delivered by Aerosol in Healthy Adult Volunteers
Acronym: COVAXAER01
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Imperial College London (Other)
Collaborators: University of Oxford (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20HH6296
Record Dates: First submitted 2021-08-12; First posted 2021-08-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: Vaccine; Vaccination; COVID-19; SARS-CoV-2; Pandemic; Immune system; Immune response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a Phase I, open label non-randomised dose escalation study in healthy adults aged 30-55 years recruited in the UK. AZD1222 will be administered by inhalation via vibrating mesh nebuliser. The study will assess safety and immunogenicity of AZD1222 with blood and respiratory tract samples. The dose evaluation will be conducted in a single centre supervised by the Chief Investigator and senior clinician experienced in first-in human studies in a cohort of 30 individuals. Approximately 14 days before vaccination, participants will undergo bronchoscopy to sample their lower airways, obtaining bronchoalveolar lavage (BAL), bronchial lining fluid and bronchial tissue. This will be repeated at day +21 and day +182 post-vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm, dose escalation (Experimental): Experimental: Healthy Volunteers Biological/Vaccine: AZD1222 (1x10^9 vp, 5x10^9 vp and 1x10^10 vp)
  Interventions: Biological: 1x10^9 vp AZD1222; Biological: 5x10^9 vp AZD1222; Biological: 1x10^10 vp AZD1222

INTERVENTIONS:
Biological: 1x10^9 vp AZD1222 — A single dose of 1x 10^9 vp AZD1222
Biological: 5x10^9 vp AZD1222 — A single dose of 5x 10^9 vp AZD1222
Biological: 1x10^10 vp AZD1222 — A single dose of 1x10^10 vp AZD1222

SUMMARY:
This study will test the COVID-19 vaccine candidate AZD1222 to investigate its safety, tolerability and capability of boosting immune responses both in the blood and the lung when administered to the respiratory tract, in volunteers previously vaccinated by intramuscular COVID-19 vaccination. Using standardised methods, we will measure immune responses in the blood, nose and lower airway and compare with data from ongoing clinical trials of intramuscular vaccination. Thus, we will show the effect of the delivery method and provide the critical information required to begin further clinical trials to show the efficacy of this needle-free vaccination strategy for booster vaccination.

DETAILED DESCRIPTION:
This is a Phase I, open label non-randomised dose escalation study in healthy adults aged 30-55 years recruited in the UK. AZD1222 will be administered by inhalation via vibrating mesh nebuliser. The study will assess safety and immunogenicity of AZD1222 with blood and respiratory tract samples. The dose evaluation will be conducted in a single centre supervised by the Chief Investigator and senior clinician experienced in first-in human studies in a cohort of 30 individuals. Approximately 14 days before vaccination, participants will undergo bronchoscopy to sample their lower airways, obtaining bronchoalveolar lavage (BAL), bronchial lining fluid and bronchial tissue. This will be repeated at day +21 and day +182 post-vaccination.

The dose escalation cohort will proceed through low (1x10^9), medium (5x10^9) and high (1x10^10 vp) dose as follows: The first participant will receive the low dose and be invited to enter information on local and systemic reactions into a diary that evening and daily thereafter for 6 days. At 48 hours post-vaccination, the team will call the first participant and go through their diary. If the reactions are Grade 1-2 or transient Grade 3 that resolved within 24 hours, two further participants will receive the same dose. At 48 hours post-vaccination, the team will call participants 2 and 3 to go through their diaries.

Provided there are no safety concerns, the fourth participant can proceed to receive the medium dose. The steps above will be repeated in order to escalate to the highest dose (1x 10^10 vp). Provided there are no safety concerns outlined, a further 6 participants will be vaccinated at the maximum tolerated dose - a total of 9 individuals vaccinated with the maximum tolerated dose. The DSMB chair will review safety data before each dose escalation and the full DSMB will periodically assess safety data every 4-8 weeks and/or as required.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 30-55 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner and access all medical records when relevant to study procedures.
* For females only, willingness to practice continuous highly effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening, bronchoscopy and vaccination.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.
* Have had a complete COVID-19 vaccination course (as one or two intramuscular injections depending on the authorisation schedule) with the last injection at least 30 days before enrolment
* Sero-suitable i.e. with evidence of SARS-CoV-2 vaccine-induced antibody responses but no evidence of previous SARS-CoV-2 infection by an authorised serology test. Those with indeterminate levels and no history of laboratory-confirmed SARS-CoV-2 infection may be included or excluded at the PI's discretion on a case-by-case basis.

Exclusion Criteria:

* History of laboratory-confirmed SARS-CoV-2 infection.
* Acute upper respiratory infection (URI or sinusitis) in the past 6 weeks
* Prior receipt of any vaccine within ≤30 days prior to enrolment or planned receipt of any vaccine within 30 days after the study vaccination
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Inhaled bronchodilator or steroid use within the last 12 months
* Intranasal steroid use within the last 6 months
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids.
* Any autoimmune conditions, except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease not requiring immunosuppressive or immunomodulatory therapy.
* History of allergic disease or reactions likely to be exacerbated by any component of the AZD1222 vaccine.
* Any history of angioedema.
* Any history of anaphylaxis.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study (e.g. ongoing severe depression, history of admission to an in-patient psychiatric facility, recent suicidal ideation, history of suicide attempt, bipolar disorder, personality disorder, alcohol and drug dependency, severe eating disorder, psychosis, use of mood stabilisers or antipsychotic medication).
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
* History of frequent nose bleeds
* Any other serious chronic illness requiring hospital specialist supervision.
* Chronic respiratory diseases, including mild asthma (resolved childhood asthma is allowed)
* Smoking (includes any inhaled product, such as cigarettes and vapes) in the past 6 months OR >5 pack-year lifetime history.
* Chronic cardiovascular disease (including hypertension), gastrointestinal disease, liver disease (except Gilberts Syndrome), renal disease, endocrine disorder (including diabetes) and neurological illness (excluding migraine)
* Seriously overweight (BMI≥40 Kg/m2) or underweight (BMI≤18 Kg/m2)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 3 months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests. Grade 1 abnormalities are permissible at investigator discretion.
* Clinically relevant abnormality on chest X-ray
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* A history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia or antiphospholipid syndrome or vaccine-induced thrombosis with thrombocytopenia

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Day 0-7
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following vaccination, measured with self-reported symptoms recorded using vaccination diaries.
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Day 0-7
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following vaccination, measured with self-reported symptoms recorded using vaccination diaries.
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Day 0-28
  Occurrence of unsolicited adverse events (AEs) for 28 days following vaccination, measured with self-reported symptoms recorded using vaccination diaries and/or AEs reported post 7 days recorded in CRFs by study team.
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Screening to Day 28
  Change from baseline for safety laboratory measures, determined by blood samples drawn at enrolment (before vaccination), Day 3, 7 and 28.
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Screening to Day 364
  Occurence of SAEs reported throughout the study.
To assess the safety, tolerability and reactogenicity profile of the candidate vaccine AZD1222 delivered by aerosol | Screening to Day 364
  Occurence of SAEs of special interest reported throughout the study.

SECONDARY OUTCOMES:
To assess cellular and humoral immunogenicity of AZD1222 | Screening to Day 364
  Interferon-gamma (IFN-y) enzyme-linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein in blood
To assess cellular and humoral immunogenicity of AZD1222 | Screening to Day 364
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) in blood

OTHER OUTCOMES:
To explore the immunology of participants | Screening to Day 364
  Virus neutralising antibody (NAb) assays against live and/or pseudotype SARS-CoV-2 virus in blood
To explore the immunology of participants | Screening to Day 364
  Cell analysis by flow cytometry assays on blood and BAL
To explore the immunology of participants | Screening to Day 364
  Interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein in bronchoalveolar lavage
To explore the immunology of participants | Screening to Day 364
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) in respiratory lining fluid and saliva
To assess changes in commensal organisms in response to vaccination | Screening to Day 364
  Quantify S protein expression in bronchial mucosa following vaccine administration using confocal microscopy
Analyse immunology to assess changes in commensal organisms in response to vaccination | Screening to Day 364
  Analysis of microbiota in nasopharyngeal and/or stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Chris Chiu, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The expectation is that after analysis the data from this study will be widely distributed in the medical and scientific community. Facilitated with presentations at local, national and international meetings, the hope is to publish widely in the medical literature. In addition, there is an excellent media department at Imperial College that will publicise research that has public interest when it is published.
  The Investigators will be involved in reviewing drafts of the manuscripts, abstracts, press releases and any other publications arising from the study. Data from the study may also be used as part of a thesis for a PhD or MD.
  All data will be anonymised and aggregated or pseudonymised; no identifying participant information will be published.
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available approximately 6 months from the last patient's last visit and remain available indefinitely.
Access Criteria: According to study protocol.